CLINICAL TRIAL: NCT04503005
Title: Effect of Fasting Duration During a Time-Restricted Eating Diet Protocol
Brief Title: Fasting Time Effects in Time-Restricted Eating (FaTE-TRE)
Acronym: FaTE-TRE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Antonio Paoli, Full Professor, University of Padova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FaTE-TRE
Record Dates: First submitted 2020-07-30; First posted 2020-08-06 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Healthy Diet; Fasting, Intermittent
Keywords: time restricted eating; intermitted fasting; body composition; metabolism; inflammation
MeSH Terms: conditions — Intermittent Fasting; Inflammation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Effect of fasting duration (Active Comparator): study the effect of different daily fasting duration on body composition and blood lipid and inflammatory markers in healthy adults.
  Interventions: Other: Time Restricted Eating
- Effect of time restricted eating protocol on chronotype (Other): study the effect of 2 month of time restricted eating on the chronotype profile of healthy adults.
  Interventions: Other: Time Restricted Eating

INTERVENTIONS:
Other: Time Restricted Eating — Effect of 16, 14 or 12 hours of daily fasting

SUMMARY:
Over the past century, lifestyles and eating habits have rapidly changed, helping to increase the onset of conditions such as obesity, metabolic syndrome and the risk of cardiovascular and metabolic diseases such as diabetes.

Recently, dietary regimens such as calorie restriction and intermittent fasting have been promoted as new strategies for reducing obesity and related co-morbidities. These strategies have proven effective in reducing body fat, improving blood pressure, lipid profile and insulin resistance in overweight individuals. However, due to the rigidity of these food protocols, the adherence of subjects to the diet is often limited or maintained only for short periods.

Time-Restricted Eating (TRE) is a less extreme form of intermittent fasting, in which the subject's daily calorie intake is consumed only in a certain period of time during the day (normally 8-12 hours). TRE have been able to reduce fat mass, pro-inflammatory markers (eg IL-6, TNF-a) and have improved some biomarkers related to cardiovascular risks (eg Insulin, HDL, TG).

The literature offers numerous versions of intermittent fasting, and the role of fasting duration is not yet fully clear. Thus. the aim of the present study is to investigate the effect od different duration of fasting in a TRE protocol on body composition and lipid and inflammatory profile. Moreover, the study intended to explore the effect of 2 month of TRE on long term maintenance of diet habits, body composition, lipid and inflammatory profile.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18-30 kg/m2
* Stable body weight for at least 3 months

Exclusion Criteria:

* type 2 Diabetes or pre-diabetes for ADA guidelines
* Significant Chronic disease
* recent and acute inflammatory status
* Recent (within 3 months) treatment with anabolic steroids, systemic corticosteroids or estrogen.
* regular exercise training (≥ 2 sessions/week) or ≥ 10,000 steps/day

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Body composition | 2 months
  change of body fat percentage measured via DEXA

SECONDARY OUTCOMES:
Blood cholesterol (total, HDL, LDL) | 2 months
  Change in blood lipid profile
Blood cytokines (IL-6; IL-1, TNF-a) | 2 months
  Change in blood inflammatory markers
Morningness-Eveningness Questionnaire (MEQ) on chronotype | 6 month
  effect od diet in eating behaviours. Minimum value is 16, maximum value is 86 Morningness-Eveningness Questionnaire (MEQ) scale is 0-41, evening type; 42-58 Neither-type; 58-68 Morning-type

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Moro, Ph.D, Principal Investigator — University of Padova
Locations (1):
- Nutrition and Exercise Lab, DSB, University of Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Derived] Sampieri A, Paoli A, Spinello G, Santinello E, Moro T. Impact of daily fasting duration on body composition and cardiometabolic risk factors during a time-restricted eating protocol: a randomized controlled trial. J Transl Med. 2024 Nov 29;22(1):1086. doi: 10.1186/s12967-024-05849-6. PMID 39614235